CLINICAL TRIAL: NCT06727721
Title: Safety and Efficacy of OCN19-overexpressed Human Umbilical Cord-derived Mesenchymal Stem Cells in the Treatment of Refractory Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lu jin ，MD (Other)
Responsible Party: Sponsor-Investigator, Lu jin ，MD, Director of endocrinology Department, Changhai Hospital, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHEC2023-226
Record Dates: First submitted 2024-11-27; First posted 2024-12-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-08

CONDITIONS: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The placebo group (Placebo Comparator): The control group was given albumin
  Interventions: Biological: albumin injection
- The control group (Active Comparator): The control group was given mesenchymal stem cells
  Interventions: Biological: Mesenchymal stem cells
- The experimental group (Experimental): The experimental group was given OCN-19 stem cells
  Interventions: Biological: mesenchymal stem cells with OCN-19

INTERVENTIONS:
Biological: mesenchymal stem cells with OCN-19 — The patient received mesenchymal stem cells with OCN-19 three times
  Arms: The experimental group
Biological: Mesenchymal stem cells — Ordinary mesenchymal stem cells were given
  Arms: The control group
Biological: albumin injection — Placebo
  Arms: The placebo group

SUMMARY:
Umbilical cord mesenchymal stem cell injection expressing OCN19, while playing the role of MSCs, can directly stimulate the expression of insulin gene and the division and proliferation of islet beta cells, which is expected to further enhance the therapeutic effect of stem cells. In non-clinical studies, it was found that MSCs expressing OCN19 had better hypoglycemic effect than MSCs

ELIGIBILITY:
1. Inclusion Criteria:

   1. Accoding to WHO diagnostic standards, patients with type 2 diabetes (fasting blood glucose ≥ 7.0 mmol/L), 30-75 years old, regardless of gender;
   2. Able to clearly understand the purpose of clinical trials and comply with trial requirements, willing to participate in this study, and sign an informed consent form;
   3. 20kg/m2 ≤ Body Mass Index (BMI) ≤ 30 kg/m2;
   4. 7.5% ≤ glycated hemoglobin ≤ 10%;
   5. Insulin should be subcutaneously injected for more than six months, and insulin and/or other oral hypoglycemic drugs (limited to metformin only) should be used α The dosage of glycosidase inhibitors remained stable for the first 3 months before randomization;
   6. During the study period, all males and females with reproductive potential were willing to accept the use of efficient contraceptive methods.
2. Exclusion Criteria:

   1. 1 Type diabetes, pregnancy diabetes or other special type diabetes patients;
   2. Patients with severe allergic constitution or allergic to any ingredients used in cell culture;
   3. Patients who have used drugs that affect glucose metabolism within the past month, such as glucocorticoids, thiazide diuretics, oral contraceptives, tricyclic antidepressants, etc;
   4. Screening the patients with acute complications such as diabetes ketoacidosis and non ketotic hyperosmolar syndrome in recent 6 months;
   5. Serious cardiovascular and cerebrovascular events such as NYHA grade III or IV heart failure, myocardial infarction, cerebral infarction, and cerebral hemorrhage occurred within the past 6 months;
   6. Patients with abnormal blood routine (including white blood cell or neutrophil count below the lower limit of normal, abnormal platelet count, and hemorrhagic disease);
   7. Patients with liver and kidney dysfunction: such as serum bilirubin TBIL exceeding the upper limit of normal by 1.5 times, AST and ALT exceeding the upper limit of normal by 2.5 times, and serum creatinine exceeding 1.5 mg/dl for males and 1.4 mg/dl for females;
   8. Patients with other serious systemic diseases (such as malignant tumors, central nervous system, cardiovascular system, blood system, digestive system, endocrine system, respiratory system, urogenital system, immune system, etc.);
   9. Individuals who are currently using systemic hormones (such as glucocorticoids), immunosuppressants, or cytotoxic therapy;
   10. Patients who received antibiotic treatment within the three months prior to study registration;
   11. Patients who have received live or attenuated vaccines within 4 weeks prior to registration, or plan to receive live or attenuated vaccines during the study period;
   12. Patients who are positive for HbsAg, Anti HCV, HIV or syphilis;
   13. Patients with active infection (such as hepatitis B or hepatitis C, tuberculosis) requiring treatment;
   14. Fever related diseases of unknown origin;
   15. Disabled patients (blind, deaf, mute, intellectually disabled, physically disabled) and individuals with mental illnesses;
   16. Patients who use drugs or have a history of adverse drug abuse and alcohol dependence within 5 years (with mental or substance abuse disorders that may interfere with the requirements of the trial);
   17. Patients of childbearing age who are pregnant or lack effective contraceptive measures or have a pregnancy plan, as well as breastfeeding patients;
   18. Patients who have received other stem cell treatments or participated in other clinical studies within the first three months of screening;
   19. Patients who have not recovered due to adverse events (≥ level 2) caused by drug treatment within 4 weeks prior to the start of the study;
   20. Patients with congenital or acquired immune dysfunction or a history of organ transplantation;
   21. Patients with other serious diseases that may affect infusion results;
   22. According to the judgment of the researchers, patients whose clinical conditions are not suitable for inclusion in this study.-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2028-12-12 (Estimated); Study Completion 2029-12-12 (Estimated)

PRIMARY OUTCOMES:
Daily insulin dose is used | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment

SECONDARY OUTCOMES:
Changes in Fasting Blood Glucose Levels Over Time | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment
  Fasting Blood Glucose (FBG) Definition: Blood sugar levels measured after fasting for at least 8 hours. Methods of measurement: Blood samples are determined using standardized laboratory analytical methods.
  Unit: Expressed in mg/dL (mg/dL). Time point: Measurements were taken at baseline, 12 and 24 weeks post-treatment.
  Goal: The target fasting blood glucose level in the study was <100 mg/dL.
Concentration of Hemoglobin A1c in Participants | From enrollment to 3 months, 6 months and 1 year after treatment
  Definition: The proportion of hemoglobin bound to glucose that reflects average blood sugar levels over the past 2-3 months.
  Methods of measurement: Blood samples were analyzed using high performance liquid chromatography (HPLC).
  Unit: Expressed in percentage (%). Time point: Measurements were taken at baseline, 12 and 24 weeks post-treatment.
  Target: The target HbA1c level in the study was <7.0%.
Concentration of fasting c-peptide in Participants | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment
  Definition: Clarify the definition of fasting C-peptide, which usually refers to the level of C-peptide measured in the fasting state, C-peptide is a by-product of insulin synthesis and reflects the function of islet beta cells.
  Measurement methods: Describe specific methods used to measure C-peptide, such as enzyme-linked immunosorbent assay (ELISA) .
  Units: Usually expressed in picmole/liter (pmol/L) or nanogram/milliliter (ng/mL).
Concentration of Glycated albumin in Participants | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment
  Definition: The proportion of albumin bound to glucose, reflecting the average blood sugar level over the past 2-3 weeks.
  Methods of measurement: Blood samples were analyzed using immunoassays. Unit: Expressed in percentage (%)
Concentration of 2-hour postprandial C-peptide in Participants | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment
  Definition: 2-hour postprandial C-peptide refers to the level of C-peptide measured 2 hours after eating, C-peptide is a by-product of insulin synthesis, reflecting the function of islet beta cells and insulin secretion capacity.
  Methods of measurement: Blood samples are analyzed using standardized methods such as enzyme-linked immunosorbent assay (ELISA) or radioimmunoassay (RIA).
  Units: Usually expressed in picomoles per liter (pmol/L) or nanograms per milliliter (ng/mL).
Concentration of total cholesterol in Participants | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment
  Definition: Total cholesterol is the sum of all cholesterol in the blood, including low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), and very low-density lipoprotein cholesterol (VLDL-C). Total cholesterol level is an important indicator of cardiovascular health.
  Methods of measurement: Blood samples are tested using standardized blood chemical analysis methods, usually enzymatic or chemical.
  Unit: Usually expressed in milligrams per deciliter (mg/dL).
  Target value: The normal range of total cholesterol in the study is usually:
  Ideal level: <200 mg/dL Marginal high levels: 200-239 mg/dL High level: ≥240 mg/dL
Concentration of LDL in Participants | From enrollment to 1 month, 3 months, 6 months and 1 year after treatment
  Low Density Lipoprotein Cholesterol (LDL-C) Definition: Low-density lipoprotein cholesterol (LDL-C) is a major form of cholesterol transport in the blood and is often referred to as "bad cholesterol." High levels of LDL-C are associated with an increased risk of cardiovascular disease, atherosclerosis, and other cardiovascular events.
  Methods of measurement: Blood samples are tested using standardized blood chemical analysis methods, usually enzymatic or chemical.
  Unit: Usually expressed in milligrams per deciliter (mg/dL).
  Target values: The normal range of LDL-C in studies is usually:
  Ideal level: <100 mg/dL Near ideal/borderline high l

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes